CLINICAL TRIAL: NCT02463968
Title: A Pilot Study of the Pathogenesis of Chikungunya Arthritis in the Americas
Brief Title: Chikungunya Arthritis in the Americas
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Global Disease Research (Unknown); US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency); Broad Institute of MIT and Harvard (Other); Allied Research Society (Unknown)
Responsible Party: Principal Investigator, Aileen Chang, Assistant Professor, George Washington University
Other Study IDs: 20150352
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Chikungunya; Arthritis
MeSH Terms: conditions — Chikungunya Fever; Arthritis | interventions — Phlebotomy; Blood Specimen Collection; Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cohort 1 CHRONIC CHIKUNGUNYA: Blood samples include one cell preparation tube with Sodium Citrate will be collected for cytokine analysis by mesoscale and mass spectrophotometer analyses, one blood RNA tube for PCR and one blood DNA tube for HLA typing. Synovial fluid samples will be drawn for chronic patients with a knee effusion with one CPT and a blood RNA tube.
  Cohort 2 ACUTE CHIKUNGUNYA: Blood samples include one CPT for evaluation of biomarkers by mass spectrophotometry, two blood RNA tubes drawn for mass spectrophotometry of viral signaling and genomic analysis and one blood DNA tube for genomic analysis.
  Cohort 3 HEALTHY CONTROLS: Participants will have one blood RNA tube, one blood DNA tube, and one CPT tube drawn as controls for the other measurements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CHRONIC CHIKUNGUNYA: Twenty participants with chronic chikungunya defined as continued knee joint effusion at least three months after diagnosis of chikungunya will be enrolled in the study.
  Interventions: Procedure: Venipuncture for blood draw; Procedure: Arthrocentesis for synovial fluid draw
- ACUTE CHIKUNGUNYA: Ten participants with acute chikungunya defined as clinical symptoms of chikungunya with acute fever and joint pain within 10 days the onset of symptoms.
  Interventions: Procedure: Venipuncture for blood draw
- HEALTHY CONTROLS: Five healthy controls will have only blood drawn once.
  Interventions: Procedure: Venipuncture for blood draw

INTERVENTIONS:
Procedure: Venipuncture for blood draw — Samples will include blood. Blood samples will be collected via venipuncture.This is a part of standard of care of new new onset joint effusion and is not a novel intervention.
Procedure: Arthrocentesis for synovial fluid draw — Samples will include joint fluid analysis in participants with a knee effusion. Synovial fluid will be drawn via arthrocentesis under sterile conditions. This is a part of standard of care of new new onset joint effusion and is not a novel intervention.
  Groups: CHRONIC CHIKUNGUNYA

SUMMARY:
Chikungunya is a mosquito-borne viral illness that leads to chronic joint pain in approximately one half of patients. The mechanisms leading to long term arthritis in humans has not been well established. There is some evidence from animal studies that activated macrophages with persistent viral infection may play a role in chronic arthritis however these mechanisms have not yet been identified in humans. It is hypothesized that activated macrophages harboring persistent active chikungunya virus are responsible for chronic arthritis and joint pain in patients. The focus of this proposal is to evaluate synovial fluid and blood for direct viral persistence and activated macrophages that may clarify the mechanism of inflammatory injury. The results of this study will be directly applicable to tailoring trials of therapeutics.

DETAILED DESCRIPTION:
Chikungunya is rapidly spreading throughout the Americas and causes debilitating chronic arthritis in approximately one fourth of patients. There is currently no standard treatment for chikungunya arthritis, and the mechanisms leading to this chronic arthritis are unclear. Further characterization of the disease pathophysiology is needed in order to guide evaluation of potential therapeutics. It is hypothesized that chronic chikungunya arthritis is due to persistence of active virus in the synovial fluid where macrophages serve as a viral reservoir. The predominance of activated macrophages in persistently infected tissue and the presence of viral genome within these macrophages in non-human primates makes our hypothesis plausible. To test this hypothesis, this study has three Specific Aims. Aim 1, describe host characteristics affect susceptibility to severe or persistent arthritis. Aim 2, determine if chikungunya virus persists in synovial fluid and synovial fluid macrophages in humans as shown in non-human primates. Aim 3, investigate how these macrophages may be activated and modulated by cytokines. To date, these pathophysiologic factors have not been well characterized in humans. Information gained from this study can directly lead to recommendations for the further evaluation of antiviral versus immune modulating medications.

ELIGIBILITY:
Inclusion Criteria:

* There will be three cohorts of patients.

  * Cohort 1 Chronic chikungunya: Twenty participants with chronic chikungunya with knee effusion defined as continued knee joint effusion at least three months after diagnosis of chikungunya.
  * Cohort 2 Acute chikungunya: Ten participants with acute chikungunya defined as clinical symptoms of chikungunya with acute fever >38°C and joint pain within 10 days the onset of symptoms without other more likely diagnosis or laboratory confirmed chikungunya.
  * Cohort 3 Healthy controls: Five healthy participants will participate that will provide baseline measurements of the cytokine profile and mononuclear cell sample recovery.

All subjects will be adults ≥18 years old. Cohort 1 participants will only be enrolled in the study if they have a knee effusion at baseline presentation. Laboratory confirmation of chikungunya includes positive viral PCR or positive IgM antibody. All patients will be able to understand and give informed consent in Spanish.

Exclusion Criteria:

* Participants will be excluded if they have a known bleeding disorders or if they are on warfarin, clopidogrel, and ticagrelor therapy they will be excluded for increased bleeding risk.
* The study will also exclude children, adults unable to give consent, prisoners, and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients living in Baranquilla, Colombia during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-08-27 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Presence of chikungunya virus in the synovial fluid of chronic arthritis patients | Participants will be followed for the duration of a clinic visit which has an expected average time of 1-2 hours
  Assess the joint for persistence of the chikungunya virus

SECONDARY OUTCOMES:
Disease Severity Measured by Disease Activity Score-28 Validated Composite Measure | Participants will be followed for the duration of a clinic visit which has an expected average time of 1-2 hours
  Disease Severity Measured by Disease Activity Score-28 Validated Survey that is a series of questions about disease severity that gives a composite score for arthritis severity and C-reactive protein level measured in mg/L.
Inflammatory Cytokine Levels | Participants will be followed for the duration of a clinic visit which has an expected average time of 1-2 hours
  Inflammatory cytokines such as IL-10, IL-6, GM-CSF, TNF, IL-2, IL-4, and IL-13 in units of pg/ml will be assessed and compared between acute and chronic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Y Chang, MD MSPH, Principal Investigator — George Washington University

REFERENCES:
- [Derived] Chang AY, Martins KAO, Encinales L, Reid SP, Acuna M, Encinales C, Matranga CB, Pacheco N, Cure C, Shukla B, Ruiz Arteta T, Amdur R, Cazares LH, Gregory M, Ward MD, Porras A, Rico Mendoza A, Dong L, Kenny T, Brueggemann E, Downey LG, Kamalapathy P, Lichtenberger P, Falls O, Simon GL, Bethony JM, Firestein GS. Chikungunya Arthritis Mechanisms in the Americas: A Cross-Sectional Analysis of Chikungunya Arthritis Patients Twenty-Two Months After Infection Demonstrating No Detectable Viral Persistence in Synovial Fluid. Arthritis Rheumatol. 2018 Apr;70(4):585-593. doi: 10.1002/art.40383. Epub 2018 Mar 7. PMID 29266856